CLINICAL TRIAL: NCT07188025
Title: Adjuvant Chemotherapy for Prevention of Recurrence in Patients With Detectable ctDNA After Surgery in High-Risk Rectal Cancer
Brief Title: ctDNA-Based Adjuvant Chemotherapy for High-Risk Rectal Cancer
Acronym: REACT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Prospectief Landelijk CRC Cohort (PLCRC) (Unknown); Dutch Colorectal Cancer Group (DCCG) (Unknown)
Responsible Party: Principal Investigator, Mirthe Ubink, MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL82006.078.22; 2024-517700-12-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-03; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer
Keywords: ctDNA; Adjuvant Chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: The proposed study is conducted within the prospective Dutch ColoRectal Cancer (PLCRC) cohort and follows the trial within cohort (TwiCs) design, i.e. a randomised controlled trial within a prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Control group ctDNA+
- Adjuvant chemotherapy (Experimental): Intervention group ctDNA+
  Interventions: Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Adjuvant chemotherapy — Adjuvant chemotherapy consists of 6 cycles of 5FU/folinic acid and oxaliplatin (FOLFOX) every 2 weeks, or 4 cycles of capecitabine and oxaliplatin (CAPOX). Duration of treatment will be 3 months (12 weeks).
  Arms: Adjuvant chemotherapy

SUMMARY:
The goal of this clinical trial is to investigate whether adjuvant chemotherapy can prevent disease recurrence in patients with high-risk rectal cancer who have detectable ctDNA after surgery.

The main research question the REACT study aims to answer is:

- Does adjuvant chemotherapy improve disease-free survival in patients with high-risk rectal cancer with detectable ctDNA after surgery?

Interventions:

- Patients with detectable ctDNA after surgery and randomised to the experimental group will be offered adjuvant chemotherapy (4 cycles CAPOX/6 cycles FOLFOX) within 12 weeks after surgery.

DETAILED DESCRIPTION:
Rationale - Rectal cancer is a worldwide cause of cancer related mortality. The incidence of rectal cancer in the Netherlands is approximately 3500 patients per year. The introduction of combined neoadjuvant (chemo)radiotherapy and total mesorectal excision (TME) has significantly reduced the local recurrence rate, but distant recurrence rates remain around 30%. Recurrences are likely to derive from residual local disease or subclinical metastatic disease (minimal residual disease). These micro metastases are undetectable by the currently used imaging techniques but still present after surgery. Adjuvant chemotherapy might be beneficial for patients at high risk for recurrence. However, there are only a few randomised controlled trials on perioperative chemotherapy available. Studies on adjuvant chemotherapy in rectal cancer yielded conflicting results. As a consequence, treatment with adjuvant chemotherapy in patients with rectal cancer is not evidence based and therefore not standard of care in the Netherlands. Recent studies suggest that preoperative intensive chemotherapy with radiotherapy, compared to standard chemotherapy and radiotherapy, resulted in a prolonged disease-free survival and overall survival. However, this was at the cost of increased toxicity, and whether the observed improvement in overall survival can be attributed to the addition of neo-adjuvant intensive chemotherapy is under debate. Consequently, there is an urgent need for biomarkers to identify those patients at high risk to recur after standard treatment, to select the patients that might benefit the most from adjuvant chemotherapy.

Objective - To investigate disease-free survival in patients with high-risk rectal cancer by treating these patients with adjuvant chemotherapy in case of detectable ctDNA after surgery.

Main trial endpoints - The primary endpoint of the study will be disease-free survival in the intention-to-treat population, calculated from the date of surgery to the date of recurrence or death from any cause of the patient, whichever occurs first.

Secondary trial endpoints - Secondary outcomes will be disease-free survival, carried out as per protocol analysis to analyse pure treatment effect. In addition, overall survival will be calculated measured from the date of surgery to the date of death from any cause. Quality of life will be assessed in both groups by obtaining already completed questionnaires provided by the PLCRC cohort study to compare the effect of adjuvant chemotherapy on quality of life. The robustness of ctDNA as biomarker will be analysed by comparing the disease-free survival of patients with detectable ctDNA who are not treated adjuvant chemotherapy (control group) with patients with undetectable ctDNA. The clearance of ctDNA of the patients who received adjuvant chemotherapy in the experimental group will be compared with the patients in the control group. Lastly, the co-occurrence of ctDNA in peripheral blood at the timing of detection of recurrent disease on imaging will be studied.

Trial design - The proposed study is conducted within the prospective Dutch ColoRectal Cancer (PLCRC) cohort and follows the trial within cohort (TwiCs) design, i.e. a randomised controlled trial within a prospective cohort.

Trial population - Patients ≥ 18 years of age with primary resected rectal cancer that meet the inclusion criteria, participating in the PLCRC cohort with informed consent for randomisation and considered physically fit for adjuvant chemotherapy are eligible.

Interventions - Patients with detectable ctDNA after surgery and randomised to the experimental group will be offered adjuvant chemotherapy within 8 weeks of surgery and no longer than 12 weeks after surgery. Adjuvant chemotherapy consists of 6 cycles of 5FU/folinic acid and oxaliplatin (FOLFOX) every 2 weeks, or 4 cycles of capecitabine and oxaliplatin (CAPOX). Duration of treatment will be 3 months (12 weeks).

Ethical considerations - In current clinical practice there is no indication for adjuvant chemotherapy for patients after surgery for primary rectal cancer. Therefore, all participating patients have no indication for adjuvant chemotherapy. Patients randomised to the experimental group will be offered adjuvant chemotherapy to reduce recurrence. According to routine clinical care, patients receiving adjuvant chemotherapy will undergo blood withdrawals and visit their treating physician before every cycle of chemotherapy. The combination chemotherapy schedule of CAPOX and FOLFOX is commonly administered in the adjuvant setting in current practice for colorectal cancer, therefore the risks and toxicity of the used adjuvant chemotherapy are well-known. The majority of side-effects are manageable and transient. The risk of the withdrawal of extra tubes of blood during regular blood withdrawal in all study participants is negligible. The benefit for participants enrolled in this trial is the potential chance to reduce their risk of recurrence with adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria

* Detectable ctDNA in the postoperative blood sample
* Age ≥ 18 years
* WHO performance score 0-1
* Informed consent for PLCRC with specific consent for additional blood withdrawals and offering of future experimental research
* Informed consent for the REACT trial.
* Histological confirmed rectal cancer; either treated with neoadjuvant (chemo)radiotherapy, and/or clinical/pathological T3/T4 and/or N+ in case no neoadjuvant therapy was administered.
* Eligible to receive treatment with combination adjuvant chemotherapy (CAPOX/FOLFOX) according to the treating physician.
* Mentally competent and able to read and understand Dutch language.

Exclusion Criteria:

* Metastatic disease
* Another malignancy in previous 5 years, with the exception of treated carcinoma in situ or skin cancer other than melanoma
* Incomplete primary tumour resection (R1 or R2 resection)
* Contra-indication for fluoropyrimidines or oxaliplatin
* Neoadjuvant oxaliplatin based systemic treatment, e.g. treated with the RAPIDO regimen consisting of short course radiotherapy followed by 6 cycles of CAPOX or 9 cycles of FOLFOX prior to surgery
* Patients with a clinical complete response, who will not undergo surgery.
* Pregnant and lactating women
* History of psychiatric disability judged by the investigator to be clinically significant, precluding informed consent or interfering with compliance of the intervention group
* Serious concomitant systemic disorders that would compromise the safety of the patient or his/her ability to complete the study, at the discretion of the investigator
* Serious infections (uncontrolled or requiring treatment)
* Current or recent (within 28 days prior to randomisation) treatment with another investigational drug or participation in another study interfering with the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2030-10 (Estimated); Study Completion 2035-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival, intention-to-treat | Calculated from the date of surgery to the date of progression (recurrence) or death from any cause of the patient, whichever occurs first, assessed up to 2 years of follow-up
  To investigate whether the disease-free survival in patients with rectal cancer who have detectable ctDNA after primary tumour resection, can be improved by administration of adjuvant chemotherapy.

SECONDARY OUTCOMES:
Overall survival, intention-to-treat | From the date of surgery to the date of death from any cause of the patient, with a median follow-up of 5 years
  To investigate whether overall survival of rectal cancer patients with detectable ctDNA after surgery can be improved with adjuvant chemotherapy
Disease-free survival, per-protocol | Calculated from the date of surgery to the date of progression (recurrence) or death from any cause of the patient, assessed up to 2 years of follow-up
  To compare all (eligible) patients in the control group to patients in the experimental group who actually started the adjuvant chemotherapy by a per protocol analysis (for pure treatment effect) for disease-free survival.
Overall survival, per-protocol | Calculated from the date of surgery to the date of death from any cause of the patient, with a median follow-up of 5 years
  To compare all (eligible) patients in the control group to patients in the experimental group who actually started the adjuvant chemotherapy by a per protocol analysis (for pure treatment effect) for overall survival.
The effect of adjuvant chemotherapy on quality of life - EQ-5D-5L | Questionnaires are obtained within PLCRC at baseline, 3 months, 6 months, 1 year, 1.5 years, 2 years and yearly after, assessed up to 4 years of follow-up
  To compare the effect of adjuvant chemotherapy on quality of life - EQ-5D-5L
The effect of adjuvant chemotherapy on quality of life - QLQ-C30 | Questionnaires are obtained within PLCRC at baseline, 3 months, 6 months, 1 year, 1.5 years, 2 years and yearly after, assessed up to 4 years of follow-up
  To compare the effect of adjuvant chemotherapy on quality of life - QLQ-C30
The effect of adjuvant chemotherapy on quality of life - QLQ-CR29 | Questionnaires are obtained within PLCRC at baseline, 3 months, 6 months, 1 year, 1.5 years, 2 years and yearly after, assessed up to 4 years of follow-up
  To compare the effect of adjuvant chemotherapy on quality of life - QLQ-CR29
Comparing disease-free survival of patients with detectable ctDNA but without receiving adjuvant chemotherapy with patients with undetectable ctDNA | Calculated from the date of surgery to the date of progression (recurrence) or death from any cause of the patient, assessed up to 2 years of follow-up
  The disease-free survival of ctDNA negative patients will be collected and analysed to confirm the robustness of postoperative ctDNA as biomarker in rectal cancer.
Comparing overall survival of patients with detectable ctDNA but without receiving adjuvant chemotherapy with patients with undetectable ctDNA | Calculated from the date of surgery to the date of death from any cause of the patient, with a median follow-up of five years
  Overall survival of ctDNA negative patients will be collected and analysed to confirm the robustness of postoperative ctDNA as biomarker in rectal cancer.

OTHER OUTCOMES:
The proportion of ctDNA-positive patients with specific mutational profiles. | Assessed from the blood sample taken 14-28 days after rectal surgery.
  To determine the mutational profile and ctDNA levels in ctDNA-positive patients.
Correlations between ctDNA mutational profiles and clinical/pathological parameters and time to recurrence | Assessed from the blood sample taken 14-28 days after rectal surgery.
  To identify and analyse specific mutations detected in ctDNA and their correlation with clinical and pathological parameters, as well as time to recurrence.
Concordance rate (%) between mutations identified in ctDNA and matched tumour tissue | Assessed from the blood sample taken 14-28 days after rectal surgery.
  To compare the mutational status of ctDNA with the mutational profile of available tumour tissue in patients, assessing concordance and potential discrepancies.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis Verhoef, MD, PhD, Principal Investigator — Erasmus Medical Center

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT07188025/Prot_SAP_000.pdf